CLINICAL TRIAL: NCT05278897
Title: Soft Tissue Adapted Hyaluronic Acid Functional Evaluation (SAFE): A Prospective Study
Brief Title: Hyaluronic Acid for Soft Tissue Injuries
Acronym: SAFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Global Research Solutions (Industry)
Collaborators: Pendopharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2022-03-02; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Elbow Tendinopathy; Ankle Sprains
MeSH Terms: conditions — Elbow Tendinopathy; Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Soft Tissue Adapted Biocompatible Hyaluronic Acid (Experimental): Soft Tissue Adapted Biocompatible Hyaluronic Acid is a clear solution of sterile 1% sodium hyaluronate (10 mg/mL) contained in a 1.2 mL pre-filled syringe. Patients will receive two injections, spaced 2 to 3 days apart (for ankle sprains) or 7 days apart (for elbow injections).
  Interventions: Device: Soft Tissue Adapted Biocompatible Hyaluronic Acid

INTERVENTIONS:
Device: Soft Tissue Adapted Biocompatible Hyaluronic Acid — 1% sodium hyaluronate

SUMMARY:
Soft Tissue Adapted Biocompatible Hyaluronic Acid, or STABHA™, has demonstrated varying degrees efficacy in patients treated for common musculoskeletal tendinopathies and ligament injuries, such as ankle sprains, lateral elbow tendinopathy, and rotator cuff tendinopathies. Factors associated with prognosis following treatment remain largely unknown. Identifying appropriate patient populations for use of STABHA™ is a necessary first step to facilitate the design of future clinical trials in the management of acute and chronic musculoskeletal soft-tissue injuries.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older.
2. Having a STABHA™ injection for the treatment of:

   1. Acute first or second degree ankle sprain (e.g. occurred within the past 48 hours).
   2. Lateral epicondylitis (tennis elbow).
3. Informed consent obtained.

Exclusion Criteria:

1. Medical contraindication to STABHA™.
2. Previous treatment with STABHA™.
3. Ankle or foot fracture.
4. Bilateral ankle sprain.
5. Previous ankle sprain in the past 12 months.
6. Prior surgical management of the ankle or elbow.
7. Current or anticipated incarceration.
8. Terminal illness with expected survival less than 90 days.
9. Currently enrolled in a study that does not permit co-enrollment.
10. Unable to obtain informed consent due to language barriers.
11. Unable to comply with the protocol.
12. Problems, in the judgment of study personnel, with maintaining follow-up with the patient.
13. Prior enrollment in the study.
14. Other reason to exclude the patient, as approved by the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-14 (Estimated); Primary Completion 2024-05-13 (Estimated); Study Completion 2024-05-13 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Pain | 12 months
  A 100mm visual analog scale, with 0 representing no pain and 100 representing the worst pain imaginable. The patient will place an 'X' on the line which represents their current pain.

SECONDARY OUTCOMES:
EuroQol-5 Dimensions (EQ-5D) | 12 months
  A quality-of-life measurement instrument based on 5 dimensions of quality of life: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. This brief questionnaire determines a quality of life score between 0 and 1, where 1 represents perfect health and 0 represents death.
12-Item Short Form Survey Version 1 (SF-12V1) | 12 months
  The SF-12 is a validated quality-of-life measurement tool that focuses on the impact of patient health on their everyday life. The SF-12 consists of 12 items that were developed to capture the physical and mental aspects of the patient's health status and is measured on a scale of -, with higher scores indicating better physical and mental health of the patient.
Pain medication use | 12 months
  The need for the patient to take pain medication for their injury/condition will be recorded using a 4-point Likert scale in order to determine if the treatment can reduce or cease the need for pain medication from medication use at baseline.
Adverse Events | 12 months
  Any adverse event experienced by the patient will be recorded at all follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, Principal Investigator — Global Research Solutions